CLINICAL TRIAL: NCT01494389
Title: The Role of CD4+T Lymphocyte Subsets in Cell Immunity in Patients With Sepsis
Brief Title: The Changes of CD4+T Lymphocyte Subsets in Septic Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chinese PLA General Hospital (Other)
Other Study IDs: 20111013-008
Record Dates: First submitted 2011-12-16; First posted 2011-12-19 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-07

CONDITIONS: Sepsis; SIRS(Systemic Inflammatory Response Syndrome)
Keywords: CD4+T lymphocyte subsets; sepsis; immunoparalysis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- SIRS: (1) temperature > 38oC or < 36oC; (2) pulse rate > 90 beats/min; (3) ventilation rate > 20 breaths/min or hyperventilation with a partial pressure of arterial carbon dioxide (PaCO2) < 32 mmHg; (4) white blood cell (WBC) count >1 2,000μL-1 or < 4000 μL-1 , or > 10% immature cells.
- sepsis: SIRS + infection
- Normal: not SIRS and have no infection

SUMMARY:
The purpose of this study is to explore the value of CD4+T lymphocyte subsets in cell immunity in the patients with sepsis.There are immunoparalysis in septic patients,the important player is the change of CD4+T lymphocyte,this immunoparalysis state contribute to the illness progress and outcome. Comprehend the change regularity of septic patients' cell immunity can guide fiter and correcter treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged 18 years old and over;
* Fulfilled at least two criteria of systemic inflammatory response syndrome (a) core temperature higher than 38 °C or lower than 36 °C (b)respiratory rate above 20/min, or PCO2 below 32 mmHg (c) pulse rate above 90/min, and (d) white blood cell count greater than 12,000/μl or lower than < 4,000/μl or less than 10% of bands.
* Clinically suspected infection;

Exclusion Criteria:

* were under 18 years of age;
* were refused by the patients or his/her familiality;
* were suffering from acquired immunodeficiency syndrome,virlhepatitis,autoimmune diseases and hematology;
* use medicine which can affect immune system,such as Glucocorticoid and Immunosuppressant
* died within 24h after being taken into the ICU, or refused to get involved in the study, or gave up treatment during the period of observation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects were selected from among inpatients who were hospitalized between March 2010 and March 2011 in the Respiratory ICU, Surgical ICU, and Emergency ICU, Chinese People's Liberation Army (CPLA) General Hospital.
Sampling Method: Non-Probability Sample
Dates: Start 2011-08; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Xie Li Xin, Doctor, Study Director — Department Of Respiratory Diseases, Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China